CLINICAL TRIAL: NCT01666990
Title: Phase 1/2 Study of Tripterygium Wilfordii Hook F (TwHF) Treatment for Evaluation the Efficacy and Safety in Immune Non-responders With HIV-1 Infection
Brief Title: Tripterygium Wilfordii Hook F (TwHF) Treatment for Immune Non-responders With HIV-1 Infection
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Beijing302-007
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Human Immunodeficiency Virus
Keywords: Tripterygium wilfordii Hook F (TwHF); HIV; CD4; immune over-activation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TwHF, lifestyle counseling (Experimental): Participants will receive TwHF (20mg each time, 3 times per day, for 48 weeks) from Day 0 through the Week 48 study visit.
  Interventions: Drug: TwHF
- placebo, Lifestyle (Placebo Comparator): Participants will receive placebo treatment (20mg each time, three times per day for 48 weeks) from Day 0 through the Week 48 study visit.
  Interventions: Drug: placebo treatment

INTERVENTIONS:
Drug: TwHF — Taken oral, three times per day, at a dose of 20 mg/time for 48 weeks.
  Other Names: treatment
  Arms: TwHF, lifestyle counseling
Drug: placebo treatment — Taken oral, three times per day, at a dose of 20 mg/time for 48 weeks.
  Other Names: placebo
  Arms: placebo, Lifestyle

SUMMARY:
HIV-1 infection is characterized by progressive depletion of CD4+ T cells that eventually leads to clinically significant immunodeficiency. A chronic generalized immune activation is now being recognized to be the main driving force for T cell depletion, loss of anti-HIV-1 immunity and disease progression during chronic HIV-1 infection. However, it is still unknown whether reducing immune activation will restore CD4 T cell counts and leading to immune reconstitution in chronic HIV infection. Tripterygium Wilfordii Hook F (TwHF) has been demonstrated to decrease immune activation of the host, and can suppress inflammation in human diseases. Here, the investigators propose a hypothesis that TwHF can reduce immune over-activation which subsequently leads to the restoration of CD4 T-cell counts and immune reconstitution in HIV-infected immune non-responders.

DETAILED DESCRIPTION:
Although HIV-1 infection is characterized by progressive depletion of CD4+ T cells that eventually leads to clinically significant immunodeficiency, a chronic generalized immune activation is now being recognized to be the main driving force for T cell depletion, loss of anti-HIV-1 immunity and disease progression during chronic HIV-1 infection. In particular, this immune activation has been identified as a disease determinant independent of viral load or cell death in HIV-1 infection. A series of clinical evidences have indicated that activated CD8 T cells may attack body cells infected with viruses. Because of this, CD4 cells infected with HIV are frequently destroyed by CD8 cells.

In traditional Chinese medicine, extracts of the roots of the medicinal vine Tripterygium wilfordii Hook F (TwHF) (known in China as "lei gong teng" or "thunder god vine") have shown therapeutic promise in treating autoimmune and inflammatory conditions as well as cancer. In this extracts, three diterpenoids-triptolide, tripdiolide, and triptonide-are the most abundant and account for the immunosuppressive and anti-inflammatory effects observed in both in vitro and in vivo studies. Recently, different extracts of TwHF have been used in Chinese allopathic medicine for the treatment of autoimmune and inflammatory diseases, and small controlled trials reported good responses with TwHF extracts in patients with cadaveric kidney transplants and Crohn disease. In particular, a multicenter, double-blind, active comparator trial of a standardized TwHF extract in patients with active rheumatoid arthritis has shown a 20% improvement in American College of Rheumatology criteria in patients with TwHF than with sulfasalazine. Thus, TwHF may reduce inflammatory responses and promote tissue recovery in human diseases.

The purpose of this study is to learn whether and how well TwHF reduces the level of activation of CD8 cells in people infected with HIV. The decreased activation of CD8 cells may lead to a more CD4 T cell restoration and immune reconstitution in HIV infection. This study will also look at how well TwHF is tolerated and its safety in HIV- infected patients.

Participants in this study will be randomly assigned to one of two treatment arms:

Arm A: Participants will receive 48 weeks of TwHF treatment. Arm B: Participants will receive 48 weeks of placebo Study treatment will be given 20 mg, three times per day for a full 48 weeks. After treatment has started, participants will be asked to come to the clinic on Weeks 4, 8, 12, 16, 24, 36, and 48. At each visit participants will receive enough study treatment to last until the next visit. Each visit will last between 2 and 3 hours. At most visits participants will have a physical exam, answer questions about any medications they are taking and how they are feeling, and have blood drawn for safety to assess CD4/CD8 cell counts and viral load. Some additional blood will also be stored for immunology testing. At some visits participants will be asked questions about their medication and medical history, have pupils dilated, have a hearing test, and have an electrocardiogram (EKG). Some visits will require participants to arrive fasting. Pregnancy tests may also be conducted if the participant is able to become pregnant or if pregnancy is suspected.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infected
2. antiretroviral therapy (ART) for at least 24 months prior to study entry and continue within the 12 months after study entry
3. CD4 count less than or equal to 250 cells/mm3 continuously before entry and at screening, obtained within 30 days prior to study entry
4. Viral load less than or equal to 400 copies/mL obtained within 30 days prior to study entry
5. Certain specified laboratory values obtained within 30 days prior to study entry. More information on this criterion can be found in the study protocol.
6. Documentation that pre-entry specimen for the primary immune activation endpoint responses has been obtained
7. No history of CDC category C AIDS-related opportunistic infections
8. Karnofsky performance score greater than or equal to 70 within 30 days prior to study entry
9. Ability and willingness to provide informed consent

Exclusion Criteria:

1. Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to study entry
2. Renal insufficiency, defined as serum creatinine greater than 1.5 mg/L, within 30 days prior to study entry
3. History of retinal disease
4. History of neoplasm other than localized squamous cell carcinoma of the skin
5. History of cardiac conduction abnormality or cardiomyopathy. More information on this criterion can be found in the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the total CD4 T cell counts compared with CD4 T cell counts at baseline | At Baseline and at week 4, 8, 12, 24, 36 and 48

SECONDARY OUTCOMES:
the CD38 expression on CD8 T cells | At Baseline and at week 4, 8, 12, 24, 36 and 48
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | at baseline and up to week 48
plasma RNA copies/mL | At Entry and at week 12 , 24 and 48
the ratio of CD4 and CD8 T cells | At baseline and at week 4, 8, 12, 24, 36 and 48
the total cell counts of peripheral CD3 T cells | At baseline and at week 4, 8, 12, 24, 36 and 48
the total cell counts of peripheral CD45RA+CCR7+ naive T cells | At baseline and at week 4, 8, 12, 24, 36 and 48
the cytokine levels of IL-1b in the plasma | At entry and at week 12, 24 and 48
the IL-2-producing T-cell number under stimulation with HIV Gag peptide pool | At entry and at week 12, 24 and 48
the HLA-DR expression on CD8 T cells | At Baseline and at week 4, 8, 12, 24, 36 and 48
the total cell number of peripheral CD8 T cells | At baseline and at week 4, 8, 12, 24, 36 and 48
the total cell counts of peripheral CD45RA+CCR7- central memory T cells | At baseline and at week 4, 8, 12, 24, 36 and 48
the total cell counts of peripheral CD45RA-CCR7- effector memory T cells | At baseline and at week 4, 8, 12, 24, 36 and 48
the cytokine levels of IL-6 in the plasma | At entry and at week 12, 24 and 48
the cytokine levels of TNF-a in the plasma | At entry and at week 12, 24 and 48
the levels of total IgG in the plasma | At entry and at week 12, 24 and 48
the cytokine levels of IFNa in the plasma | At entry and at week 12, 24 and 48
the IFN-g-producing T-cell number under stimulation with HIV Gag peptide pool | At entry and at week 12, 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, Professor, Principal Investigator — Beijing 302 Hospital
Locations (2):
- China (2):
  - Beijing 302 Hospital, Beijing, Beijing Municipality
  - the Yunnan Hospital of Infectious Diseases, Kunming, Yunnan

REFERENCES:
- [Background] Hammer SM, Squires KE, Hughes MD, Grimes JM, Demeter LM, Currier JS, Eron JJ Jr, Feinberg JE, Balfour HH Jr, Deyton LR, Chodakewitz JA, Fischl MA. A controlled trial of two nucleoside analogues plus indinavir in persons with human immunodeficiency virus infection and CD4 cell counts of 200 per cubic millimeter or less. AIDS Clinical Trials Group 320 Study Team. N Engl J Med. 1997 Sep 11;337(11):725-33. doi: 10.1056/NEJM199709113371101. PMID 9287227
- [Background] Mocroft A, Vella S, Benfield TL, Chiesi A, Miller V, Gargalianos P, d'Arminio Monforte A, Yust I, Bruun JN, Phillips AN, Lundgren JD. Changing patterns of mortality across Europe in patients infected with HIV-1. EuroSIDA Study Group. Lancet. 1998 Nov 28;352(9142):1725-30. doi: 10.1016/s0140-6736(98)03201-2. PMID 9848347
- [Background] Appay V, Sauce D. Immune activation and inflammation in HIV-1 infection: causes and consequences. J Pathol. 2008 Jan;214(2):231-41. doi: 10.1002/path.2276. PMID 18161758
- [Background] Li T, Wu N, Dai Y, Qiu Z, Han Y, Xie J, Zhu T, Li Y. Reduced thymic output is a major mechanism of immune reconstitution failure in HIV-infected patients after long-term antiretroviral therapy. Clin Infect Dis. 2011 Nov;53(9):944-51. doi: 10.1093/cid/cir552. Epub 2011 Sep 29. PMID 21960716
- [Background] Goldbach-Mansky R, Wilson M, Fleischmann R, Olsen N, Silverfield J, Kempf P, Kivitz A, Sherrer Y, Pucino F, Csako G, Costello R, Pham TH, Snyder C, van der Heijde D, Tao X, Wesley R, Lipsky PE. Comparison of Tripterygium wilfordii Hook F versus sulfasalazine in the treatment of rheumatoid arthritis: a randomized trial. Ann Intern Med. 2009 Aug 18;151(4):229-40, W49-51. doi: 10.7326/0003-4819-151-4-200908180-00005. PMID 19687490
- [Background] Kupchan SM, Court WA, Dailey RG Jr, Gilmore CJ, Bryan RF. Triptolide and tripdiolide, novel antileukemic diterpenoid triepoxides from Tripterygium wilfordii. J Am Chem Soc. 1972 Oct 4;94(20):7194-5. doi: 10.1021/ja00775a078. No abstract available. PMID 5072337
- [Background] Ji SM, Wang QW, Chen JS, Sha GZ, Liu ZH, Li LS. Clinical trial of Tripterygium Wilfordii Hook F. in human kidney transplantation in China. Transplant Proc. 2006 Jun;38(5):1274-9. doi: 10.1016/j.transproceed.2006.03.017. PMID 16797280
- [Background] Tao X, Lipsky PE. The Chinese anti-inflammatory and immunosuppressive herbal remedy Tripterygium wilfordii Hook F. Rheum Dis Clin North Am. 2000 Feb;26(1):29-50, viii. doi: 10.1016/s0889-857x(05)70118-6. PMID 10680192
- [Background] Qiu D, Zhao G, Aoki Y, Shi L, Uyei A, Nazarian S, Ng JC, Kao PN. Immunosuppressant PG490 (triptolide) inhibits T-cell interleukin-2 expression at the level of purine-box/nuclear factor of activated T-cells and NF-kappaB transcriptional activation. J Biol Chem. 1999 May 7;274(19):13443-50. doi: 10.1074/jbc.274.19.13443. PMID 10224109
- [Background] Tao X, Schulze-Koops H, Ma L, Cai J, Mao Y, Lipsky PE. Effects of Tripterygium wilfordii hook F extracts on induction of cyclooxygenase 2 activity and prostaglandin E2 production. Arthritis Rheum. 1998 Jan;41(1):130-8. doi: 10.1002/1529-0131(199801)41:13.0.CO;2-4. PMID 9433878